CLINICAL TRIAL: NCT03238053
Title: Laser Treatment of Genito-urinary Syndrome in Women With Breast and Endometrial Cancer and Menopausal Women
Brief Title: Laser Treatment of Genito-urinary Syndrome in Women
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Hospital terminated treatment with laser
Sponsor: Herning Hospital (Other)
Responsible Party: Principal Investigator, Finn Lauszus, Senior Consultant, Research Specialist, Herning Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Laser treatment
Record Dates: First submitted 2017-08-01; First posted 2017-08-03 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Laser-Induced Scar; Breast Cancer; Endometrial Cancer; Menopause; Vaginal Atrophy; Bladder, Overactive
Keywords: laser treatment, randomized trial, menopause, vaginitis, urge
MeSH Terms: conditions — Breast Neoplasms; Endometrial Neoplasms; Urinary Bladder, Overactive; Vaginitis

STUDY DESIGN:
Intervention Model Description: Four Groups of women randomized for thre months to either laser og sham treatment
Who Masked: Participant
Masking Description: Laser probe perform similar noise and movement without providing rays
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Menopausal Laser (Active Comparator): 20 women with vaginal laser treatment
  Interventions: Procedure: Vaginal laser treatment; Device: laser system
- Menopausal sham (Sham Comparator): 20 women with probe, no active laser ray
  Interventions: Device: sham
- breast cancer laser (Active Comparator): 20 women with breast cancer with vaginal laser treatment
  Interventions: Procedure: Vaginal laser treatment; Device: laser system
- breast cancer sham (Sham Comparator): 20 women with breast cancer with vaginal probe, no active laser rays
  Interventions: Device: sham
- endometrial cancer laser (Active Comparator): 20 women with endometrial cancer with vaginal laser treatment
  Interventions: Procedure: Vaginal laser treatment; Device: laser system
- endometrial cancer sham (Sham Comparator): 20 women with endometrial cancer with vaginal probe, no active laser rays
  Interventions: Device: sham
- overactive bladder laser (Active Comparator): 20 women with overactive bladder with vaginal laser treatment
  Interventions: Procedure: Vaginal laser treatment; Device: laser system
- Overactive bladder sham (Sham Comparator): 20 women with overactive bladder with vaginal probe, no active laser rays
  Interventions: Device: sham

INTERVENTIONS:
Procedure: Vaginal laser treatment — Fractional CO 2 laser system (SmartXide 2 V 2 LR,DEKA, Florence, Italy), using the following setting: dot power 30 watt, dwell time 1000 μ s, dot spacing 1000 μ m and the smart stack parameter from 1 to 3. The laser beam is provided using a vaginal probe, which is gently inserted up to the top of the vaginal canal and subsequently withdrawn and rotated in order to provide a complete treatment of the vaginal wall. At the level of the vaginal introitus, the dot power is decreased to 20 watt 27 . A treatment cycle includes three laser applications (every 4 weeks). The procedure is performed in the outpatient clinic and does not require any specific preparation (e.g. analgesia/anesthesia).
  Arms: Menopausal Laser; breast cancer laser; endometrial cancer laser; overactive bladder laser
Device: sham — Fractional CO 2 laser system (SmartXide 2 V 2 LR,DEKA, Florence, Italy), using the following setting: dot power 30 watt, dwell time 1000 μ s, dot spacing 1000 μ m and the smart stack parameter from 1 to 3. The laser beam is provided using a vaginal probe, which is gently inserted up to the top of the vaginal canal and subsequently withdrawn and rotated in order to provide a complete treatment of the vaginal wall. At the level of the vaginal introitus, the dot power is decreased to 20 watt 27 . A treatment cycle includes three laser applications (every 4 weeks). The procedure is performed in the outpatient clinic and does not require any specific preparation (e.g. analgesia/anesthesia).
  Arms: Menopausal sham; Overactive bladder sham; breast cancer sham; endometrial cancer sham
Device: laser system — FractionalCO 2 laser system (SmartXide 2 V 2 LR,DEKA, Florence, Italy), using the following setting: dot power 30 watt, dwell time 1000 μ s, dot spacing 1000 μ m and the smart stack parameter from 1 to 3. The laser beam is provided using a vaginal probe, which is gently inserted up to the top of the vaginal canal and subsequently withdrawn and rotated in order to provide a complete treatment of the vaginal wall. At the level of the vaginal introitus, the dot power is decreased to 20 watt 27 . A treatment cycle includes three laser applications (every 4 weeks). The procedure is performed in the outpatient clinic and does not require any specific preparation (e.g. analgesia/anesthesia).
  Arms: Menopausal Laser; breast cancer laser; endometrial cancer laser; overactive bladder laser

SUMMARY:
Women with genitourinary syndrome of menopause, overactive bladder, with breast or endometrial cancer are randomized to either laser treatment og sham treatment for 3 months. The randomization is stratified for estrogen treatment. The effect is evaluated by questionnaire, histology and microbiology swaps

DETAILED DESCRIPTION:
Genitourinary syndrome of menopause (GSM) is characterized by symptoms such as vaginal dryness, dyspareunia, irritation, urinary incontinence, overactive bladder , and urinary tract infections. GSM replaces the previous term vulvovaginal atrophy as agreed upon by a joint terminology conference sponsored by the North American Menopause Society and the International Society for the Study of Women's Sexual Health. GSM is a new terminology more accurate than the terms of VVA/atrophic vaginitis, because it describes the clinical signs and symptoms of the vulva, vagina and lower urinary system. In contrast, VVA/atrophic vaginitis describes the appearance of the vulvovaginal structures only. The GSM has a prevalence of more or less 50%, depending on country of origin, with a negative impact on sexuality, quality of life and well-being.

The aging process is genetically determined and environmentally modulated. Estrogen deficiency occurring after menopause causes a series of modifications in many different areas of the female body, including the pelvic floor. Menopause can, therefore, lead to functional genital or urinary symptoms impacting women's quality of life. It is debatable to which extent modifications and symptoms occurring after menopause are related to estrogen deficiency or to the aging process per se. Vulvovaginal atrophy (VVA) involves histological, morphological, microbiological, and clinical changes. These include alteration in collagens, decreased quantity of elastic fibers, reduced vascularization, thinning and flattening of the vaginal epithelium, and production of glycogen, an essential factor for the growth of vaginal lactobacilli. As a consequence, the vaginal canal becomes shorter and narrower, and the vaginal epithelium becomes paler and more likely to develop petechiae. Further, a decrease in Lactobacillus species and a rise of vaginal pH values over 4.5 are observed, resulting in the loss of the local vaginal defense mechanisms against bacterial pathogens, which may predispose to local inflammation and/or infections.

Women with VVA commonly complain of vaginal dryness, burning, irritation or itching, and dyspareunia. Local estrogens represent the first-line therapy for VVA. However, women's compliance with and preference for this treatment are poor; alternatives and palliative solutions, such as moisturizing or lubricant local creams or gels, are commonly proposed. In recent years, fractional CO 2 laser has become a popular, efficient, precise, and safe system, particularly for dermatologists and plastic surgeons. CO 2 laser has many applications, including treatment of skin lesions (ie, seborrheic keratosis, syringomas, and xanthelasmas around the eye), warts, and toenail diseases, as well as anti-aging function.

Various therapeutic strategies, hormonal or not, oral or local, have been proposed for the improvement of the vaginal microecosystem of postmenopausal women (e.g. estrogens, probiotics, combination of vaginal estrogens with live Lactobacillus). Hormonal therapy (oral or local) has been associated with a healthier vaginal microecosystem by repopulating the Lactobacillus species to a premenopausal status and by reducing the pH of vaginal fluid.

In women treated for estrogen dependent cancer i.e. endometrial and breast cancer women and practioners are reluctant to use estrogens and favor non-hormonal treatment modalities. The effect of these on the histological, microbiological and clinical symptoms is poorly understood and lack randomized trials to evaluate effect. Several proof of concept and feasibility studies have shown clinical effects of laser as potential treatment but little is known if it can stand alone or if supplementation with estrogens may benefit the clinical symptoms and vulvovaginal environment further. Thus, the ideal management for the achievement of the optimal benefit - risk balance is still under investigation. The choice of treatment is often guided by clinical experience and patient preference.

In postmenopausal women, the disturbance of Lactobacillary flora was correlated with the presence of Gardnerella vaginalis, Trichomonas vaginalis, enterococci, group B streptococci, and Escherichia coli. Available data indicate that pre-existing vaginal colonization with pathogenic enterobacteria is essential for the appearance and recurrence of urinary tract infections (UTIs). Indeed, postmenopausal women are prone to UTIs with an incidence of about 8% per year and a 4% likelihood of recurrence, while symptomatic bacteriuria was estimated in up to 15% of women. The general population of lactobacilli, as assessed in the routine practice, provides indirect information regarding the estrogenic status. To our knowledge there is currently no evidence regarding the potential impact that the intravaginal laser therapy may have on the vaginal microenvironment in women with symptoms of GSM.

Laser treatment improves significantly the VVA symptoms, sexual function and quality of life of postmenopausal women, as well as the vaginal health index. Other studies found restored thickness of the squamous stratified epithelium of the vaginal mucosa with a significant storage of glycogen in the epithelial cells and remodelling the vaginal connective tissue with the production of new collagen and ground substance molecules.

Breast cancer is the most common cancer in women in Denmark, annually ca. 4600 women are diagnosed with the disease, of whom 30% are under the age of 55. Most patients undergo breast conserving surgery followed by adjuvant therapy. Adjuvant therapy varies according to stage of disease, but radiotherapy is often added, as well as chemotherapy. If the cancer is hormonally responsive, long term antihormonal treatment is also given, such as the selective estrogen receptor modulator (SERM) tamoxifen for pre-menopausal women, that works as a inhibitor of estrogen in breast tissue, but as an estrogen in other tissues such as the endometrium. Post-menopausal women with hormone responsive breast cancer are treated with aromatase inhibitors for five years. Most side effects associated with tamoxifen (TAM) and aromatase inhibitors (AIs) are related to estrogen deprivation, and the symptoms are similar to those experienced during natural menopause. It has been reported that up to 50-75% of breast cancer survivors experience one or more genitourinary symptoms and puts the sexual life of women under stress. Postmenopausal women may have many common age-related symptoms but also have the above mentioned iatrogenic factors entering their lives to aggravate the symptom complex.

The aim of the current study was to assess the effect of laser laser therapy with and without local estrogens. The study groups consist of 1) postmenopausal women and 2 ) women treated for breast cancer. The laser treatment was given randomized to these women. The effects were evaluated in the histopathology of the vagina, the vaginal microenvironment, and health related questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* menopause i.e. age more than 50 years and absence of menstruation for twelve months
* breast cancer
* endometrial cancer
* symptoms of vaginal dryness
* dyspareunia rated as moderate or severe most bothersome symptoms

Exclusion Criteria:

* use of vaginal moisturizers, lubricants or any other local preparation within the thirty days prior to inclusion
* acute or recurrent urinary tract infections
* active genital infections i.e. herpes genitalis, candida
* previous reconstructive pelvic surgery
* pelvis organ prolapse stage 2
* any serious disease or chronic condition that could interfere with study compliance except from breast and endometrial cancer
* psychiatric disorders precluding informed consent

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Visual analogue score on vaginal symptoms | three months
  10-cm VAS to measure the overall satisfaction with vaginal symptoms, where the left extreme of the scale indicated ' the worst level of satisfaction ' and the right indicated ' the best level of satisfaction

SECONDARY OUTCOMES:
histopathology | three months
  Qualitative analysis of the microscopic and ultrastructural aspects of the collagenic and elastic components of the matrix is performed. A specific image analysis with computerized morphometry is performed to demonstrate the specific action of CO2 laser and possibly to correlate the modifications of the ultrastructural pattern with specific molecular modifications. We also consider the fine cytological aspects of connective tissue proper cells, particularly fibroblasts, under the conditions of the specific laser stimulation.
microbiology | three months
  a sterile swab is inserted into the vaginal canal and a sample obtained from the posterior fornix of the vagina. Vaginal samples are placed in a transport gel (Stuart). pH indicator strips (MColorpHastTM, Merck, Germany) are applied against the lateral vaginal wall using sterile forceps, followed by a vaginal lavage for wet mount. Smears from vaginal samples are placed on a glass slide, observed under microscope for Trichomonas vaginalis and Candida species and stained afterwards according to standard Gram stain procedure. Cultures for aerobic and anaerobic bacteria species are performed, using MacConkey agar, blood agar, Sabouraud dextrose agar, chocolate agar as culture media, focusing on bacteria with potential clinical impact (e.g. aerobic vaginitis39, UTIs, vaginal candidiasis).

CONTACTS AND LOCATIONS:
Overall Officials: Sine Jakobsen, MD, PhD, Principal Investigator — Randers Regional Hospital; Finn F Lauszus, Study Chair — Herning Hopsital
Locations (1):
- Gynecology Dept. Herning Hospital, Herning, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Salvatore S, Nappi RE, Parma M, Chionna R, Lagona F, Zerbinati N, Ferrero S, Origoni M, Candiani M, Leone Roberti Maggiore U. Sexual function after fractional microablative CO(2) laser in women with vulvovaginal atrophy. Climacteric. 2015 Apr;18(2):219-25. doi: 10.3109/13697137.2014.975197. Epub 2014 Dec 16. PMID 25333211
- [Background] Salvatore S, Leone Roberti Maggiore U, Athanasiou S, Origoni M, Candiani M, Calligaro A, Zerbinati N. Histological study on the effects of microablative fractional CO2 laser on atrophic vaginal tissue: an ex vivo study. Menopause. 2015 Aug;22(8):845-9. doi: 10.1097/GME.0000000000000401. PMID 25608269
- [Background] Athanasiou S, Pitsouni E, Antonopoulou S, Zacharakis D, Salvatore S, Falagas ME, Grigoriadis T. The effect of microablative fractional CO2 laser on vaginal flora of postmenopausal women. Climacteric. 2016 Oct;19(5):512-8. doi: 10.1080/13697137.2016.1212006. Epub 2016 Aug 24. PMID 27558459
- [Derived] Ippolito GM, Crescenze IM, Sitto H, Palanjian RR, Raza D, Barboglio Romo P, Wallace SA, Orozco Leal G, Clemens JQ, Dahm P, Gupta P. Vaginal lasers for treating stress urinary incontinence in women. Cochrane Database Syst Rev. 2025 Jul 25;7(7):CD013643. doi: 10.1002/14651858.CD013643.pub2. PMID 40709601